CLINICAL TRIAL: NCT01492842
Title: Behavioral, Immunologic and Virologic Correlates of Oral Human Papillomavirus Infection in Adolescents and Young Adults With Behaviorally Acquired HIV-Infection
Brief Title: Correlates of Oral Human Papillomavirus Infection in Adolescents and Young Adults With Behaviorally Acquired HIV
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 114
Record Dates: First submitted 2011-10-17; First posted 2011-12-15 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Youth with behaviorally-acquired HIV who enrolled in ATN 106: Behaviorally-acquired HIV-infected adolescents and young adults, ages 12-24, inclusive, who have enrolled in ATN 106.

SUMMARY:
The proposed study is a substudy of ATN 106 and a cross sectional study intended to be conducted at each of the AMTUs newly participating in ATN III. The intent is to enroll all youth with behaviorally-acquired HIV who have enrolled in ATN 106. The study involves a review of the subjects' medical chart and a collection of an oral rinse sample.

DETAILED DESCRIPTION:
ATN 114 is a cross-sectional substudy of ATN 106. In addition to sharing data collected in ATN 106, an oral rinse sample along with the subject's self reported history and medical chart abstraction of HPV vaccination status and medical chart abstraction of a history of oral condylomata, oral dysplasia and oral tumor viruses will be collected in ATN 114.

Recruitment is expected to last approximately one year, similar to the same timeframe for ATN 106. Enrollment may be terminated earlier at the discretion of the ATN Executive Committee and/or the ATN 114 protocol team should ATN 106 also terminate enrollment early. Individuals who have agreed to participate in ATN 106 may be simultaneously approached at any clinic visit, or, for community-based sites, contacted directly for participation in ATN 114. Site staff may also contact individuals via phone, e-mail, or any other agreed-upon methods of communication. Site staff should try as much as possible to incorporate the study visit into a regularly scheduled clinic visit.

ELIGIBILITY:
Inclusion Criteria

* Behaviorally acquired HIV-infection as indicated by medical chart abstraction or self-reported history of sexual risk and/or needle using behaviors; and
* Completion of the ATN 106 study visit (the same day or up to a maximum of 14 calendar days).

Exclusion Criteria

* Presence of serious psychiatric symptoms (e.g., active hallucinations, thought disorder) that would impair the individual's ability to complete the study measures;
* Visibly distraught (e.g., suicidal, homicidal, exhibiting violent behavior); or
* Intoxicated or under the influence of alcohol or other substances at the time of consent/assent for ATN 114.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Behaviorally-acquired HIV-infected adolescents and young adults, ages 12-24, inclusive, who have enrolled in ATN 106.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of HPV infection, outcome defined as HPV positive or HPV negative | 1 year
  Beta-globin positive samples (reported as Positive/negative; there is no unit of measure) will be considered evaluable and classified as HPV-positive if any of the 37 HPV DNA types were detected) and HPV negative if all HPV types were negative.

SECONDARY OUTCOMES:
Behavioral Factors | 1 year
  Sexual behaviors:
  • Sexual encounters for male/female: type of sexual contact/in the last 3 months N number of partners by type of sexual contact/in last 3 months
  Substance use behaviors:
  * Tobacco product use (ever used, frequency of use past 3 months); <= 1/month >=1/=week
  * Alcohol use (ever used, frequency of use past 3 months); Irregular/regular
  * Marijuana use (ever used, frequency of use past 3 months); <= 1/month >=1/=week
  * Cocaine use ((ever used, frequency of use past 3 months); <= 1/month >=1/=
Immunologic factors | 1 year
  The immunological factors will include CD4+ cell count (cell/uL) and severity of disease according to the CDC Staging/Immunologic Category for HIV Disease (No unit of measurements)
Virologic factors | 1 year
  HIV viral load (copies/ml), EBV [(copies of EBV PHC( per human cells)] and KSHV (HHV-8) [copies of HHV-8 PHC (per human cells)]

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kahn, MD, Study Chair — Cincinnati Childrens Hospital Medical Center
Locations (5):
- United States (5):
  - University of Colorado Denver, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - The Fenway Institute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- See also: ATN website — http://www.atnonline.org